CLINICAL TRIAL: NCT04752488
Title: The Effect of Telerehabilitation and Conventional Rehabilitation on Clinical Results and Exercise Adherence in Patients With Chronic Neck Pain
Brief Title: The Effect of Telerehabilitation in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Fatih ÖZDEN, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mugla Training and Research
Record Dates: First submitted 2021-02-10; First posted 2021-02-12 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Neck Pain
Keywords: Telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (TR) Group (Experimental): The TR group will be followed up through the video-based exercise software within the 8-week home exercise program.
  Interventions: Other: Telerehabilitation (TR)
- Conventional Rehabilitation (CR) Group (Active Comparator): The CR group will be trained face-to-face with conventional methods before the 8-week home exercise program, and an exercise program will be prescribed with a visual information form.
  Interventions: Other: Conventional Rehabilitation (CR)

INTERVENTIONS:
Other: Telerehabilitation (TR) — The home exercise program will be educated to the patient on the first day. Exercises for isometric and isotonic strengthening, stretching, and stabilization of the neck muscles will be given. Exercises will be presented to the patients in audio-video format and detailed instructions with explanations. The exercise protocol will also be the same as in the conventional rehabilitation group. Patients will be asked to do the exercises once a day for 8 weeks and 10 repetitions each.
  Arms: Telerehabilitation (TR) Group
Other: Conventional Rehabilitation (CR) — The home exercise program will be educated to the patient on the first day. Isometric and isotonic strengthening, stretching and stabilization exercises for the neck muscles will be given. Exercise information form including explanation and picture of the exercises will be given to the patients. Patients will be asked to do the exercises once a day for 8 weeks and 10 repetitions each.
  Arms: Conventional Rehabilitation (CR) Group

SUMMARY:
Telerehabilitation offers more efficient follow-up of patients during their home exercise period as a cost-effective and effective treatment model. This study was planned to examine the effectiveness of telerehabilitation in patients with chronic neck pain. The aim of the study is to compare the video-based and telerehabilitation based home-exercise program in patients with chronic neck pain. It is aimed to evaluate the patients in terms of pain, functionality, quality of life, and exercise adherence.

DETAILED DESCRIPTION:
With telerehabilitation, patients can easily adapt to home exercise programs and be monitored remotely. In this way, it will be ensured that individuals can apply their exercises at an optimum level in non-clinical settings and to prevent exercise application errors that occur due to the learning effect frequently observed in conventional methods. Exercise is considered a central element in physical therapy and rehabilitation management in patients with chronic neck pain. However, studies have found that improvements after physical therapy and rehabilitation are not preserved in the long term, and recurrence of chronic low back pain is common. With a more cost-effective treatment model, "telerehabilitation", it is aimed that patients can be followed more efficiently during their home exercise period. The aim of the study is to compare the video-based and telerehabilitation based home-exercise program in patients with chronic neck pain. It is aimed to evaluate the patients in terms of pain, functionality, quality of life, and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 - 65
* Patients who have suffered from neck pain for at least 3 months
* Signing the consent form

Exclusion Criteria:

* Situations that prevent the evaluation or communication with the individual
* Illiterate individuals
* Individuals who have undergone an operation due to neck pain problem, diagnosed with a tumor, infection, ankylosing spondylitis, rheumatoid arthritis or inflammatory diseases, fracture, cauda equina syndrome
* Conditions in which specific pathological condition is proven such as malignant condition, fracture, systemic rheumatoid disease
* Orthopedic and neurological problems that prevent evaluation and/or treatment
* Complaints of pain and numbness spreading to the upper extremities
* Individuals with a diagnosed psychiatric disease
* Individuals who have received physiotherapy in the last 6 months
* Individuals using another treatment method during the study
* Individuals with musculoskeletal pain in any other part of the body during work
* Pregnant participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 minutes
  The patients will be asked to mark their pain feelings for rest and activity on a 10 cm numerical line (0: no pain, 10: unbearable pain). It is planned to use numerical VAS in our study. The cut-off values for chronic musculoskeletal pain will be classified as the severity of pain according to VAS as follows:
  <3.4 centimeters: mild pain, 3.5-7.4 centimeters: moderate pain, > 7.5 centimeters: severe pain.
Neck Disability Index (NDI) | 5 minutes
  NDI consists of 10 titles: pain intensity, personal care, lifting, reading, headache, concentration, study, driving, sleeping, and recreation. For each item included in the study; 0 indicates "no disability" and 5 represents "complete disability" Participants will be asked to give points between these scores. The total score ranges between 0 (no disability) and 50 (complete disability).
Short Form-36 (SF-36) | 5 minutes
  SF-36 consists of thirty-six items. These provide measurements of eight dimensions. Subscales evaluate health between 0-100 points; '0' indicates poor health, '100' indicates good health.
Tampa Scale for Kinesiophobia | 5 minutes
  The scale is a 17-item. A 4-point Likert scoring (1= strongly disagree, 4= totally agree) is used in the scale. The participant gets a total score between 17-68. The high score obtained by the participant indicates that the kinesiophobia is also high.

SECONDARY OUTCOMES:
Exercise Adherence Rating Scale (EARS) | 5 minutes
  EARS provides a measurement of commitment to home exercise. This may facilitate the evaluation of interventions that promote self-management, for the treatment of chronic conditions.
Telemedicine Patient Questionnaire | 5 minutes
  Telemedicine Patient Questionnaire evaluates the usability and satisfaction of the patients. The total score is scored between 17 and 85. Higher scores indicate expectation, satisfaction and usability.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Özkeskin, PhD, Study Director — Ege University; İsmet Tümtürk, MSc, Principal Investigator — Ege University; Cem Yalın Kılınç, Principal Investigator — Muğla Sıtkı Koçman University; Fatih Özden, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No